CLINICAL TRIAL: NCT01154569
Title: Absorption of Drugs Post-Bariatric Surgery (Absorb-Azithromycin)
Acronym: Absorb-Azithro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Raj Padwal Associate Professor, Internal Medicine, University of Alberta
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0002390
Record Dates: First submitted 2010-06-21; First posted 2010-07-01 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Bariatric Surgery
Keywords: drug absorption; azithromycin; obesity; bariatric surgery
MeSH Terms: conditions — Obesity | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Post Roux-en-Y gastric bypass (Active Comparator): Post-bypass receiving a single dose of azithromycin
  Interventions: Drug: Azithromycin
- Controls (Active Comparator): BMI and sex matched. Have not undergone surgery
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — 500 mg single dose
  Other Names: Zithromax

SUMMARY:
Bariatric (obesity) surgery has become the preferred treatment option for patients with severe obesity and is increasing in popularity. It is commonly performed, with nearly 350 000 operations in the world every year. The most common type of bariatric surgery is gastric bypass, in which stomach size is reduced by 95% and the upper intestine is bypassed. Bypass of the upper intestine may lead to medication malabsorption, although this potential adverse effect has received little study.

The objective of this study is to determine whether gastric bypass reduces the absorption of a azithromycin, a medication commonly prescribed first-line for infections, especially pneumonia. Patients and non-surgical controls will receive a single dose of azithromycin under highly standardized study conditions. The absorption of azithromycin will be calculated and compared between surgical and non-surgical study groups.

The investigators hypothesis is that there will be a significant reduction in the absorption of azithromycin in gastric bypass patients compared to non-surgical controls. This raises the possibility that post-gastric bypass patients treated with azithromycin may fail to respond to treatment, become worse and even die. This study will have important implications for the large number of past and future gastric bypass recipients.

DETAILED DESCRIPTION:
In the past decade, bariatric surgery has emerged as the preferred treatment option for patients with either severe obesity [body mass index (BMI) ≥ 40 kg/m2] or moderate obesity (BMI 35.0-39.9 kg/m2) and a major medical complication (e.g., diabetes, hypertension, sleep apnea). Surgery reduces weight by 33% after 2-3 years, and is associated with improvements in obesity-related comorbidities, mortality and quality of life.

Consequently, demand for bariatric surgery is increasing at an exponential rate in Canada, the United States and globally, with 350 000 estimated surgeries performed annually globally. Laparoscopic Roux-en-Y gastric bypass is the most commonly performed type of bariatric procedure. This operation restricts stomach capacity 5% of its original size and bypasses the duodenum and much of the jejunum. The major adverse consequence of intestinal bypass is nutrient malabsorption leading to deficiencies of iron, fat-soluble vitamins and vitamin B12. The malabsorption of drugs, many of which are designed to be maximally absorbed in the upper small intestine, is also a major potential concern. Surprisingly, this issue has received surprisingly little attention in the published literature. A number of factors may contributed to reduced absorption post-bypass, delayed gastric emptying, reduced intestinal transit time, diminished opportunity for mucosal exposure, and changes in drug solubility resulting from alterations in intestinal pH.

Azithromycin, a macrolide antibiotic that interferes with ribosomal protein synthesis, is indicated for the treatment of respiratory tract, skin/soft tissue, sinus and pelvic infections. Azithromycin is most commonly prescribed orally for the treatment of community-acquired pneumonia (CAP), and is recommended as first-line treatment in patients with this condition who are being managed on an outpatient basis. CAP accounts for over 1 million physician visits, 60 000 hospital admissions, 640 000 days of restricted activity and (together with influenza) is the 6th leading cause of death in the United States. In Edmonton, at least 50% of CAP is managed as with outpatient therapy. Post-bariatric surgery patients who develop CAP and are treated with outpatient oral antibiotics would clearly be at risk of treatment failure if the antibiotic is not optimally absorbed. Treatment failure may pose a significant risk of respiratory complications or death. Unfortunately, no studies have examined the absorption of antibiotics post-gastric bypass. Because, azithromycin is intrinsically poorly absorbed, with a bioavailability of only 38%, suboptimal absorption post-gastric bypass is a major concern. The purpose of this study is to determine whether gastric bypass results in clinically significant reductions in azithromycin absorption.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female
2. 18 - 60 years old
3. ≥ 3 months post-RYGB surgery or a suitable control for bariatric surgery
4. Able to provide written informed consent.

Exclusion Criteria:

1. Undergone or undergoing reversal of a previous bariatric procedure which involves further resection or bypass of the intestine.
2. Any major post-operative gastrointestinal complications, such as an anastomotic leak, outlet obstruction or persistent vomiting
3. Currently on azithromycin therapy
4. Any contraindications to azithromycin therapy such as:

   * Allergy or hypersensitivity to the drug
   * liver failure or baseline liver enzymes higher than 3-fold above the upper limit of normal
   * end-stage renal failure (glomerular filtration rate < 10 ml/min)
   * macrolide hypersensitivity
   * history of torsade de pointes or baseline QTc interval ≥ 500 ms
   * acute illness
5. Pregnant or nursing
6. Concomitant treatment with septra, anti-HIV drugs, digoxin, disopyramide, ergotamine, dihydroergotamine, triazolam, antihistamines (terfenadine, astemizole) and theophylline is also a contraindication to enrolment because of the potential for drug interactions that would affect the blood concentrations of azithromycin or these agents.
7. Any other medical, social or geographic condition, which, in the opinion of the investigator would not allow safe completion of the study protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Azithromycin absorption | Blood samples for analysis of azithromycin levels collected at 0, 0.5, 1, 1.5, 2, 3, 5, 7 and 24 hours post-dose.
  Area-under-the-curve azithromycin absorption from 0 to 24 hours post dose.

SECONDARY OUTCOMES:
Tmax | instant
  Time to peak concentration
Cmax | instant
  Maximal concentration post-ingestion of azithromycin

CONTACTS AND LOCATIONS:
Overall Officials: Raj Padwal, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada